CLINICAL TRIAL: NCT00860639
Title: Randomized Open Phase III Trial Testing Efficacy of Gemtuzumab Ozogamycin (MYLOTARG) Associated to Intensive Chemotherapy for Patients Aged Between 18-60 Years and Presenting an Acute Myeloid Leukemia (AML) With Intermediate Risk
Brief Title: Efficacy of Gemtuzumab Ozogamycin for Patients Presenting an Acute Myeloid Leukemia (AML) With Intermediate Risk
Acronym: LAM2006IR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Chugai Pharmaceutical (Industry); French Innovative Leukemia Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/06/10-I
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; gemtuzumab ozogamycin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gemtuzumab ozogamycin (Active Comparator): Initial randomization will be completed upon receipt of karyotype results and will determine the administration of gemtuzumab ozogamycin (MYLOTARG ®) in combination with chemotherapy during the induction course and the first intensive consolidation course.
  Interventions: Drug: gemtuzumab ozogamycin
- without Mylotarg (No Intervention)

INTERVENTIONS:
Drug: gemtuzumab ozogamycin — gemtuzumab ozogamycin = 6mg/m² during the induction course (Day 4) gemtuzumab ozogamycin = 6mg/m² during the first intensive consolidation course (Day 4)
  Other Names: gemtuzumab ozogamycin (MYLOTARG ®)
  Arms: gemtuzumab ozogamycin

SUMMARY:
The main objective of the study is to improve outcome of younger patients (between 18-60 years) with acute myeloid leukemia and intermediate risk defined by the cytogenetics. In this population, in the absence of bone marrow transplantation, event free survival (EFS) is estimated at 35% after three years of follow-up. Adjunction of gemtuzumab ozogamycin (MYLOTARG®) to standard chemotherapy is supposed to increase EFS up to 50% at 3 years. To test this hypothesis, the Groupe Ouest Est d'Etude des Leucémies et Autres Maladies du Sang (GOELAMS ) sponsored by Nantes University Hospital leads this randomized open phase III trial in 29 French centers.

DETAILED DESCRIPTION:
Initial randomization will be completed upon receipt of karyotype results and will determine the administration of gemtuzumab ozogamycin (MYLOTARG ®) in combination with chemotherapy during the induction course and the first intensive consolidation course. The induction course include: Daunorubicin for 3 days (60mg/m²) associated with cytarabine (200mg/m²) for 7 days. The MYLOTARG ® will be administered according to the randomization arm on the 4th day of treatment by slow intravenous infusion of 2 hours at a dose of 6 mg/m2. Early bone marrow assessment will be performed at D15. In case of blast excess (>5%) , a second course of induction will be administered.

The consolidation treatment depends on age, molecular prognostic factors, and donor availability:

* Patients with good molecular prognosis profile [ NPM1 + / FLT3 ITD - or CEBPa mutated ] will be consolidated by two courses of intensive chemotherapy comprising Mitoxanthrone and intermediate dose of Cytarabine with or without MYLOTARG ® according to the initial randomization during the first course.
* Patients younger than 51 years, eligible for standard allogeneic transplantation with sibling or full matched unrelated donor will receive a standard bone marrow transplantation which not begin before 90 days after the induction.
* Patients with no donor or older than 50 years, or with a donor being identified, will receive two courses of intensive consolidation comprising Mitoxantrone and intermediate-dose of Cytarabine with or without Mylotarg ® 6 mg / m² during the first consolidation according to the randomisation arm.
* Patients aged 51 to 60 years with an HLA identical donor (sibling or unrelated), will receive a non-myeloablative haematopoietic stem cells transplant (HSCT) after the second course of consolidation.
* For other patients, an autologous hematopoietic stem cells transplant (HSCT) will be performed after the 2nd course of consolidation. Collection of peripheral blood stem cells (PBSCs) will be performed after the first consolidation course and a second collection may be considered after the second consolidation course in case of inadequate collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with de novo AML and intermediate risk as defined by the cytogenetics criteria of GOELAMS Group:

  * Normal karyotype or
  * Karyotype with other abnormalities, excluding the favourable group [t (15; 17), t (8; 21), inv (16)] and the high risk group [(-5/5q-, -7/7q- , t (9.22), t (6.9), 11q23 anomaly excluding the t (9; 11), abnormal 3q, complex karyotype (> 3 abnormalities)]. Not previously treated for AML.
* Patients aged 18 to 60 years
* And having more than 20% of blast cells in bone marrow and as previously described.
* And with intermediate cytogenetics as previously defined
* And whose expression of the CD33 antigen on the blasts was defined using standard method
* And with a WBC <or equal to 100G/L.
* And who can receive either one or the other of the treatments under study
* And having a good performance status (WHO score <3) with a life expectancy greater than one month.
* Affiliated with the Social Security

Exclusion Criteria:

* Patients aged under 18 or over 60 years
* OR with AML:

  * Not classifiable in the classification French-American-British (FAB)
  * Type M3
  * Or blastic transformation of a myeloproliferative or myelodysplastic syndrome previously diagnosed
  * Outside the intermediate cytogenetic group as previously defined
* OR with isolated extramedullary localization of their disease
* OR WBC> 100G / L
* Patients with known human immunodeficiency virus (HIV) infection or human T-lymphotrophic virus 1 (HTLV-1)
* Patients with SGOT/SGPT >5N
* Patients with a calculated creatinine clearance of <50 mL/min
* Informed consent refusal
* Pregnant and/or lactating female

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 327 (Actual)
Dates: Start 2007-10; Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

PRIMARY OUTCOMES:
event free survival (EFS)after 3 years for patients not eligible for standard allogenic transplantation | 3 years

SECONDARY OUTCOMES:
Complete Remission Rate (CR) Overall Survival at 3 years Relapse rate at 3 years Toxicity and tolerability of each treatment arm Evaluation of Minimal residual disease by WT1 and NPM1 study at different phases of treatment. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Delaunay, MD, Principal Investigator — Nantes University Hospital
Locations (29):
- France (29):
  - CH Pays d'Aix, Aix
  - CHU Amiens, Amiens
  - CHRU Angers, Angers
  - CH Avignon, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU Hôpital Minjoz, Besançon
  - CHU Morvan, Brest
  - CHU Hôtel Dieu, Clermont-Ferrand
  - CH Louis Pasteur, Colmar
  - CHU du Bocage, Dijon
  - CHU Michallon, Grenoble
  - CHU Dupuytren, Limoges
  - Institut Paoli Calmette, Marseille
  - CH Metz Thionvile, Metz
  - CHU Lapeyronie, Montpellier
  - CH Muller, Mulhouse
  - CHU Hôtel Dieu, Nantes
  - CHU Carémeau, Nîmes
  - CH La Source, Orléans
  - Hopital Cochin (AP-HP), Paris
  - CHU du Haut Lévèque, Pessac
  - CHU Jean Bernard - La Milétrie, Poitiers
  - CHU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - Institut de Cancérologie de la Loire, Saint-Etienne
  - CHU Hautepierre, Strasbourg
  - CHU Purpan, Toulouse
  - CHU Bretonneau, Tours
  - CHU Brabois, Vandœuvre-lès-Nancy